CLINICAL TRIAL: NCT00061633
Title: A Phase 2, Randomized, Double-Blind, Multinational Trial of Intravenous Telavancin Versus Standard Therapy for Treatment of Complicated Gram Positive Skin and Skin Structure Infections (Gram Positive cSSSI)
Brief Title: Phase 2 Trial of TD 6424 (Telavancin) Versus Standard Therapy for Complicated Gram Positive Skin and Skin Structure Infections (Gram Positive cSSSI)
Acronym: FAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I6424-202a
Record Dates: First submitted 2003-05-30; First posted 2003-06-02 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Infections, Gram-Positive Bacterial; Abscess; Burns; Cellulitis; Ulcer; Wound Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Abscess; Burns; Cellulitis; Ulcer; Wound Infection | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Standard of care for cSSSI (Active Comparator): cSSSI - complicated skin and skin structure infections
  Interventions: Drug: Vancomycin or antistaphylococcal penicillin

INTERVENTIONS:
Drug: Telavancin — Telavancin 7.5 mg/kg/day IV (intravenously) for up to 14 days
  Other Names: VIBATIV; TD-6424
  Arms: Telavancin
Drug: Vancomycin or antistaphylococcal penicillin — Vancomycin 1 Gram IV (intravenously) every 12 hrs or nafcillin 2 Grams, oxacillin 2 Grams, or (in South Africa) cloxacillin 0.5 - 1 Gram, IV (intravenously) every 6 hrs for up to 14 days.
  Arms: Standard of care for cSSSI

SUMMARY:
Serious infections caused by resistant bacteria are becoming more of a medical problem throughout the world. One of the ways to deal with this problem is to develop new drugs that can control these bacteria. This study will measure how well TD-6424 (Telavancin) can control infections and whether this drug can be safely given to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following complicated skin and skin structure infections with either a suspected or confirmed Gram positive organism as the major cause of the infection:

  * major abscess requiring surgical incision and drainage
  * infected burn (see exclusion criteria for important qualifications)
  * deep/extensive cellulitis
  * infected ulcer (see exclusion criteria for important qualifications)
  * wound infections
* Patients must be expected to require at least 4 days of intravenous antibiotic treatment

Exclusion Criteria:

* Previous systemic antibacterial therapy (with the exception of aztreonam and metronidazole) for > 24 hours within 7 days prior to the first dose of study medication unless the pathogen was resistant to prior treatment or the patient was a treatment failure (no clinical improvement after 3 days).
* Burns involving > 20% of body surface area or third degree/full thickness in nature, diabetic foot ulcers, ischemic ulcers/wounds, necrotizing fasciitis, gas gangrene, or mediastinitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2003-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- eStudy Site, 3450 Bonita Road, Ste 201, Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 05Jun03 to 20Jan04
Groups:
- Telavancin: Patients with complicated Gram-positive skin and skin structure infections were randomized to receive telavancin 10 mg/kg/day IV (intravenously)
- Standard of Care for cSSSI: Patients with complicated Gram-positive skin and skin structure infections were randomized to receive standard therapy, defined as vancomycin 1 Gram every 12 hours IV (intravenously) or an antistaphylococcal (semisynthetic) penicillin.
Period: Overall Study
Arm/Group | Telavancin | Standard of Care for cSSSI
Started | 84 | 85
Completed | 79 | 74
Not Completed | 5 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Other | 1 | 1
Not completed — Never received study treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Standard of Care for cSSSI | Total
Number analyzed (Participants) | 84 | 83 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 78 | 158
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.9) | 44.3 (13.5) | 44.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 54 | 46 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 68 | 72 | 140
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 11
  Black or African American | 21 | 20 | 41
  White | 38 | 41 | 79
  More than one race | 13 | 14 | 27
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 117
  South Africa | 25 | 25 | 50
Diabetes Status [Number; unit: participants]
  Diabetic | 25 | 19 | 44
  Non-Diabetic | 59 | 64 | 123

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Which is Measured at Test of Cure (TOC) in the Clinically Evaluable (CE) Population
Description: * Cure: Resolution of clinically significant signs, symptoms associated with the skin infection present at study admission or improvement to the extent that the infectious process had been controlled and no further therapy with study medication was necessary.
  * Failure: Inadequate response to study therapy or the need for significant surgical management (e.g. more than just routine debridement) of the infection site following antibiotic therapy and prior to the Test-of-Cure (TOC) visit.
  * Indeterminate: Inability to determine outcome.
Time Frame: 7-14 days following end of antibiotic treatment
Population: The CE population were a subset of the All Treated Population and was composed of patients who met the inclusion/exclusion criteria or were granted permission to enroll and had a clinical response of "cure" or "failure." The All Treated Population patients received at least one treatment. The Primary Efficacy Analysis was of the CE population.
Measure: Number; unit: participants
Arm/Group | Telavancin | Standard of Care for cSSSI
Number analyzed (Participants) | 72 | 69
participants
  Cured | 66 | 66
  Failure | 6 | 3
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Telavancin vs Standard of Care for cSSSI; 95% Confidence Interval: -0.1349 to 0.0485 No est. value. Parameter that was estimated: Risk Difference; Test type: Non-Inferiority or Equivalence — Sample size was selected on the basis of clinical judgment and was deemed adequate to provide clinically meaningful descriptive results consistent with study objectives. This sample size was estimated to provide 39% power to test televancin's non-inferiority to vancomycin with respect to clinical response using a non-inferiority margin of 10%; p = 0.5289, 2-sided 95% confidence interval

ADVERSE EVENTS:
Description: The Safety Population was the "All Treated Population" - all patients who received one treatment. The Primary Analysis was of the Clinically Evaluable (CE) Population. The CE population was composed of the patients who met the inclusion / exclusion criteria or were granted permission to enroll and had a clinical response of "cure" or "failure".
Arm/Group | Telavancin | Standard of Care for cSSSI
Serious Adverse Events (participants affected / at risk) | 3/84 | 9/83
Other Adverse Events (participants affected / at risk) | 46/84 | 50/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=84) | Standard of Care for cSSSI (N=83)
Cellulitis (Infections and infestations) | 0 | 3
Necrotizing Fasciitis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Wound Abscess (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Gangrene (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=84) | Standard of Care for cSSSI (N=83)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Keratoconjunctivitis Sicca (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphasia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 11
Post-Procedural Nausea (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 3
Anasarca (General disorders) | 1 | 0
Catheter related complication (General disorders) | 0 | 1
Catheter Site Inflammation (General disorders) | 1 | 0
Catheter site rash (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Feeling hot (General disorders) | 2 | 1
Feeling jittery (General disorders) | 0 | 1
Infusion site pain (General disorders) | 1 | 1
Injection Site Extravasation (General disorders) | 0 | 1
Injection site phlebitis (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pain exacerbated (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Red Man Syndrome (General disorders) | 0 | 3
Rigors (General disorders) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 0 | 3
Gonorrhea (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Localized Infection (Infections and infestations) | 1 | 0
Nasal abscess (Infections and infestations) | 0 | 1
Necrotizing Fasciitis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 1 | 1
Tinea Pedis (Injury, poisoning and procedural complications) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 4
Vaginal Candidiasis (Infections and infestations) | 1 | 0
Wound Abscess (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Blister (Injury, poisoning and procedural complications) | 1 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase increased (Investigations) | 0 | 4
Aspartate Aminotransferase increased (Investigations) | 1 | 6
Blood Alkaline phosphatase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood in stool (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 3
Blood pressure increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Hepatic Enzyme increased (Investigations) | 0 | 1
HIV Test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burning sensation (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 9 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 6 | 2
Confusional State (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Euphoric Mood (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4
Irritability (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1
Diabetic neuropathy (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Microalbuminuria (Renal and urinary disorders) | 4 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Genital Pruritis Female (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Crackles Lung (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Gangrene (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less